CLINICAL TRIAL: NCT05235100
Title: Preoperative Intensity-modulated Radiotherapy (IMRT) With Concurrent Apatinib Mesylate for Localised Extremity or Trunk Sarcoma
Brief Title: Preoperative IMRT With Concurrent Apatinib for Localised Extremity or Trunk Sarcoma （SPARE-02）
Acronym: SPARE-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principle Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-007196
Record Dates: First submitted 2021-12-02; First posted 2022-02-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma,Soft Tissue; Extremity; Trunk; Intensity-modulated Radiotherapy; Targetd Therapy; Major Wound Complications
MeSH Terms: conditions — Sarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib arm (Experimental): Apatinib 500mg QD, used 2 weeks prior to IMRT, concurrent with pre-operative IMRT, and 1 month after end of IMRT
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib Mesylate 500mg QD, begin from 2 weeks prior to IMRT, to 1 month after end of IMRT

SUMMARY:
To investigate the safety and efficacy of preoperative IMRT and concurrent Apatinib for primary truncal or extremity soft tissue sarcoma; To investigate the Quality of life and extremity function post-combination treatment; To study the mechanism of radio-sensitizing effects of Apatinib for primary truncal or extremity soft tissue sarcoma; To assess the relationship between the MRI imaging, pathological findings and local control.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18-yo.
* Histology proven soft tissue sarcoma of truncal or extremity, deemed appropriate for preoperative radiotherapy and conservative surgery by multidisciplinary discussion.
* ECOG 0-3
* Histology reviewed by reference pathologist
* Lesion can be assessed
* Can tolerate radiotherapy and Apatinib
* Agree contraception.
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed

Exclusion Criteria:

* No gross tumor post-resection in other center.
* Contraindications to Apatinib, including allergic to Apatinib, active bleeding, ulcer, enteric perforation, enteric obstruction, uncontrolled hypertension, Grade 3 to 4 cardiac insufficiency (per NYHA criteria), and severe hepatic or renal insufficiency (Grade 4), etc.
* Dermatofibrosarcoma protuberans(DFSP), Desmoids, etc.
* Benign histology
* Secondary cancer within 5 years (except cervical carcinoma in situ or early-stage skin basal cell carcinoma)
* STS can be cured by extensive operation alone.
* Previous irradiation to the same area
* radiological evidence of distant metastases
* Other contraindications, can't tolerate operation or other treatment needed in this study.
* Neoadjuvant chemotherapy given or planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of Major wound complications within 4 months post-surgery | 4-months post-surgery

SECONDARY OUTCOMES:
Acute and late toxicities | acute toxicities were evaluated during and 3 months after IMRT, late toxicities were evaluted after 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Patient-reported Quality of Life assessed by EORTC-QLQ-C30 questionnaire | From date of enrollment to 2 years after surgery, specifically at pre-IMRT, end of IMRT, 1 months post-IMRT, and every 3 to 6 months during follow-up up to 2 years post-surgery
  Evaluate the quality of life by patient-reported EORTC-QLQ-C30 questionnaire at different time points
Extremity function scores | From date of enrollment to 2 years after surgery, specifically at pre-IMRT, end of IMRT, 1 months post-IMRT, and every 3 to 6 months during follow-up up to 2 years post-surgery
  Evaluate the extremity function by MSTS (Musculoskeletal Tumor Rating Scale) and TESS (Toronto Extremity Salvage Score) forms at different time points
Pathological remission rate | 2 weeks after operation
  Evaluate the tumor remission rate microscopically 2 weeks after operation
Local control | 2-year
Overall survival | 2-year

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China